CLINICAL TRIAL: NCT02584816
Title: A Phase III, Multicenter, Open Label, Randomized Study of Bovine Rotavirus Pentavalent Vaccine (BRV-PV) to Evaluate Lot-To-Lot Consistency and to Investigate Potential Interference With Routine UIP Vaccinations in Healthy Infants in India.
Brief Title: Phase III Study on Rotavirus Vaccine to Evaluate Lot-to-lot Consistency and Interference With Routine UIP Immunization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ROTA: 04 / VAC-020
Record Dates: First submitted 2015-10-06; First posted 2015-10-23 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Rotavirus Gastroenteritis
Keywords: BRV-PV; Rotavirus vaccine; lot-to-lot consistency; interference with routine immunization
MeSH Terms: interventions — Poliovirus Vaccine, Oral; RIX4414 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 - BRV-PV Lot A (Experimental): BRV-PV Lot A + DPT- HepB-Hib + OPV
  Interventions: Biological: BRV-PV Lot A + DPT-HepB-Hib + OPV
- Group 2 - BRV-PV Lot B (Experimental): BRV-PV Lot B+ DPT- HepB-Hib + OPV
  Interventions: Biological: BRV-PV Lot B + DPT-HepB-Hib + OPV
- Group 3 - BRV-PV Lot C (Experimental): BRV-PV Lot C + DPT- HepB-Hib + OPV
  Interventions: Biological: BRV-PV Lot C + DPT-HepB-Hib + OPV
- Group 4 - ROTARIX (Active Comparator): ROTARIX + DPT-HepB-Hib + OPV
  Interventions: Biological: ROTARIX + DPT-HepB-Hib + OPV

INTERVENTIONS:
Biological: BRV-PV Lot A + DPT-HepB-Hib + OPV — Dose 1: 6-8 weeks, Dose 2: 10 week, Dose 3: 14 week
  Arms: Group 1 - BRV-PV Lot A
Biological: BRV-PV Lot B + DPT-HepB-Hib + OPV — Dose 1: 6-8 weeks, Dose 2: 10 week, Dose 3: 14 week
  Other Names: Live Attenuated human-bovine reassortant pentavalent rotavirus vaccine
  Arms: Group 2 - BRV-PV Lot B
Biological: BRV-PV Lot C + DPT-HepB-Hib + OPV — Dose 1: 6-8 weeks, Dose 2: 10 week, Dose 3: 14 week
  Arms: Group 3 - BRV-PV Lot C
Biological: ROTARIX + DPT-HepB-Hib + OPV — Dose 1: 6-8 weeks, Dose 2: 10 week, Dose 3: 14 week (Third dose-Placebo)
  Arms: Group 4 - ROTARIX

SUMMARY:
This is a Phase 3, open-label, randomized study to evaluate lot-to-lot consistency in the manufacture of Bovine Rotavirus Pentavalent Vaccine (BRV-PV).

DETAILED DESCRIPTION:
The study is designed to evaluate lot-to-lot consistency in the manufacturing of Rotavirus vaccine by testing the vaccine in infants in order to demonstrate equivalence in the induction of specific anti-rotavirus IgA antibodies across three production lots. The study will also examine the potential interference of vaccine with UIP vaccines that will be administered concurrently by assessing non-inferiority in the immune responses to those vaccines when administered with / without the study vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants as established by medical history and clinical examination before entering the study.
2. Age: 6-8 weeks at the time of enrollment.
3. Parental ability and willingness to provide written informed consent.
4. Parent who intends to remain in the area with the child during the study period.
5. Receipt of birth dose of Hepatitis B vaccine and OPV.

Exclusion Criteria:

1. Presence of diarrhea or vomiting in the previous 72 hours or on the day of enrollment (temporary exclusion).
2. Presence of fever on the day of enrollment (temporary exclusion).
3. Acute disease at the time of enrollment (temporary exclusion).
4. Concurrent participation in another clinical trial at any point throughout the entire timeframe for this study.
5. Presence of significant malnutrition or any systemic disorder as determined by medical history and / or physical examination which would compromise the subject's health or is likely to result in nonconformance to the protocol.
6. History of congenital abdominal disorders, intussusception, or abdominal surgery.
7. Known or suspected impairment of immunological function based on medical history and physical examination.
8. Household contact with an immunosuppressed individual or pregnant woman.
9. Prior receipt or intent to receive rotavirus and / or diphtheria, tetanus, pertussis, Haemophilus Influenzae type b, Hepatitis B vaccine (other than birth dose) or inactivated polio vaccine (IPV) during the study period and outside of the study. OPV dose received during national / subnational immunization days will be allowed.
10. A known sensitivity or allergy to any components of the study vaccine.
11. Clinically detectable congenital or genetic defect.
12. History of persistent diarrhea (defined as diarrhea that lasts 14 days or longer).
13. Receipt of any immunoglobulin therapy and / or blood products since birth or planned administration during the study period.
14. History of chronic administration (defined as more than 14 days) of immunosuppressants including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study.
15. History of any neurologic disorders or seizures.
16. Any medical condition in the parents / infant which, in the judgment of the Investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parents' ability to give written informed consent.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1500 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Rotavirus vaccine lots Immunogenicity | Four weeks after the third dose of vaccination
  Serum anti- rotavirus IgA antibody concentrations expressed as GMCs for the BRV-PV to demonstrate equivalence in lot consistency among three lots.
Immunogenicity of UIP vaccines | Four weeks after the third dose of vaccination

SECONDARY OUTCOMES:
Immediate adverse events and Solicited post -vaccination reactogenicity | AEs within 30 minutes post-vaccination and post vacc reactogenicity during 7 days after each vaccination
Rotavirus Immunogenicity: | Four weeks after the third dose of vaccination
  Serum anti- rotavirus IgA antibody concentrations expressed as GMCs and proportion of subjects with post-vaccination IgA antibody concentration ≥20 U/ml for the comparison of BRV-PV vaccine and licensed rotavirus vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Prasad Kulkarni, M.D., Study Director — Serum Institute of India Pvt. Ltd.
Locations (10):
- India (10):
  - Gandhi Medical College and Gandhi Hospital, Hyderabad, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - JSS Medical College and Hospital, Mysore, Karnataka
  - T. N. Medical College and B. Y. L. Nair Charitable, Mumbai, Maharashtra
  - Seth G S Medical College & KEM Hospital, Mumbai, Maharashtra
  - Bharati Vidyapeeth Medical College and Hospital, Pune, Maharashtra
  - KEM Hospital and Research Centre, Vadu, Pune, Maharashtra
  - Sri Ramachandra Medical Centre, Chennai, Tamil Nadu
  - Institute of Child Health, Kolkata, West Bengal
  - Maulana Azad Medical College, New Delhi

REFERENCES:
- [Result] Desai S, Rathi N, Kawade A, Venkatramanan P, Kundu R, Lalwani SK, Dubey AP, Venkateswara Rao J, Narayanappa D, Ghildiyal R, Gogtay NJ, Venugopal P, Palkar S, Munshi R, Bavdekar A, Juvekar S, Ganguly N, Niyogi P, Uttam KG, Kondekar A, Kumbhar D, Mohanlal S, Agarwal MC, Shetty P, Antony K, Gunale B, Dharmadhikari A, Deshpande J, Nalavade U, Sharma D, Bansal A, Tang Y, Flores J, Kulkarni PS. Non-interference of Bovine-Human reassortant pentavalent rotavirus vaccine ROTASIIL(R) with the immunogenicity of infant vaccines in comparison with a licensed rotavirus vaccine. Vaccine. 2018 Sep 5;36(37):5519-5523. doi: 10.1016/j.vaccine.2018.07.064. Epub 2018 Aug 10. PMID 30104114
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/30104114